CLINICAL TRIAL: NCT06801600
Title: A Comparative Study Between Age-Based and Weight-Based Bupivacaine Dosing for Pediatric Spinal Anesthesia in Children Undergoing Elective Infra-Umbilical Surgeries: A Randomized Double-Blinded Controlled Trial
Brief Title: Age-Based and Weight-Based Bupivacaine Dosing for Pediatric Spinal Anesthesia for Elective Infra-Umbilical Surgeries
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kareem Mohammed Assem Nawwar, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MS-503-2024
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Spinal Anesthesia; Local Anesthetic; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight-based dosing (Active Comparator): Hyperbaric bupivacaine 0.5% dosage will be calculated and administered intrathecally as 0.4 mg/kg or 0.08 ml/kg if body weight ≤ 15 kg and 0.3 mg/kg or 0.06 ml/kg if body weight > 15 kg
  Interventions: Drug: Weight-based dosing
- Age-based dosing group (Active Comparator): Hyperbaric bupivacaine 0.5% will be administered at the dose of age divided by 5 (in ml). The age in months after the completion of a year was noted and considered as the next age if it is more than 6 months and the same age if it is ≤ 6 months.
  Interventions: Drug: Age-based dosing

INTERVENTIONS:
Drug: Weight-based dosing — Hyperbaric bupivacaine 0.5% dosage will be calculated and administered intrathecally as 0.4 mg/kg or 0.08 ml/kg if body weight ≤ 15 kg and 0.3 mg/kg or 0.06 ml/kg if body weight > 15 kg
  Arms: Weight-based dosing
Drug: Age-based dosing — Hyperbaric bupivacaine 0.5% will be administered at the dose of age divided by 5 (in ml). The age in months after the completion of a year was noted and considered as the next age if it is more than 6 months and the same age if it is ≤ 6 months.
  Arms: Age-based dosing group

SUMMARY:
Pediatric anesthesia presents distinctive challenges, particularly concerning appropriate dosage administration of local anesthetics for spinal anesthesia (SA). Spinal anesthesia in infants has been linked to a lower incidence of hypotension, hypoxia, bradycardia, and postoperative apnea in comparison to general anesthesia (GA); ensuring a high level of cardiovascular and respiratory stability.

Additionally, SA has been linked to lower operating room time, post-anesthesia care unit, hospital length of stay, corticosteroid administration, narcotic requirements, postoperative emesis, and cardiopulmonary complications in comparison to GA.

A reduction in systemic blood pressure frequently accompanies neuraxial blocks in adults, necessitating intervention. Nevertheless, spinal, caudal, or epidural blocks administered to children under six years old are not associated with any substantial alterations in blood pressure. In children aged 6 to 10, there is a linear decrease in blood pressure that will reach a plateau at approximately a 30% decrease in those beyond the age of 10. Conversely, younger children require no additional precautions.

Bupivacaine, has a narrow therapeutic index in children, and its dosing requires careful consideration to strike a balance between effective anesthesia and the risk of toxicity. The traditional method of dosing bupivacaine in pediatric spinal anesthesia is based on the child's body weight. This weight-based dosing considers the assumption that children's drug clearance correlates with their body mass. However, this approach might not account for the maturational changes in drug handling by pediatric patients or the variability in spinal column length and cerebrospinal fluid volumes, not always proportional to weight but may evolve with age.

Emerging evidence suggests that age-based dosing may be more effective. It hypothesizes that developmental pharmacokinetics, including changes in body composition, organ function, and drug-receptor differences, can influence bupivacaine metabolism and action more significantly than body mass alone. By accounting for the age-related anatomical and physiological changes, age-based dosing could result in more precise and effective anesthesia with a decreased risk of adverse outcomes.

To the authors knowledge, there is no study comparing age-based and weight-based bupivacaine dosing for pediatric spinal anesthesia in children undergoing elective infra-umbilical surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II
* Both genders
* Elective infra-umbilical surgeries with anticipated duration ≤ 90 minutes.

Exclusion Criteria:

* Guardian refusal.
* Children with major congenital heart disease, including septal defects.
* Patients with neuromuscular disorders or high intracranial pressure.
* Children with spinal deformities or morbid obesity (BMI above the 99th percentile).
* Children with a history or family history of coagulation disorders.
* Children with local infection at the site of skin puncture for spinal anesthesia.
* Children with known allergy to bupivacaine.
* Surgeries requiring head down (Trendelenburg) or prone position.
* Unexpected prolongation of surgery > 90 minutes.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
The peak sensory level | 5 mins after intrathecal bupivacaine injection
  The sensory level of subarachnoid block, tested by firm skin pinch.

SECONDARY OUTCOMES:
Block level time | 10 minutes from intrathecal injection of local anesthetic
  Time from injection of local anesthetic intrathecally to achieving full motor and adequate sensory block
Duration of the block | 120 minutes from intrathecal injection of local anesthetic
  Duration from intrathecal injection of local anesthetic till return of motor power of the lower limbs
Postoperative pain score | 3 hours from intrathecal injection of local anesthetic
  Postoperative pain levels using the Face, Legs, Activity, Cry, and Consolability (FLACC) scale
Incidence of failed spinal blocks | 2 hours from attempting subarachnoid block application
  Percentage of failed spinal blocks requiring conversion to general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Manal M Elgohary, M.D., Study Chair — Cairo University; Hany M Elhady, M.D., Study Director — Cairo University; Kareem MA Nawwar, M.D., Study Director — Cairo University; Bassant A Heikal, M.B.B.Ch., Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No